CLINICAL TRIAL: NCT04959578
Title: Comparison of Darbepoetin Alpha and Recombinant Human Erythropoietin as Erythropoietic Agents for Treatment of Anemia in Pediatric Chronic Kidney Disease Patients
Brief Title: Comparison of Darbepoetin Alpha and Recombinant Human Erythropoietin for Treatment of Anemia in Children With Chronic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rufaida Mazahir (Other)
Responsible Party: Sponsor-Investigator, Rufaida Mazahir, Principal Investigator, Sir Ganga Ram Hospital
Organization: Sir Ganga Ram Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/01/18/1317
Record Dates: First submitted 2021-07-03; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: Anemia; Chronic kidney disease; Darbepoetin alpha; Erythropoietin; Pediatric
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erythropoietin (Active Comparator): Recombinant Human Erythropoietin
  Interventions: Drug: Recombinant human erythropoietin
- Darbepoetin alfa (Experimental): Darbepoetin Alpha
  Interventions: Drug: Darbepoetin Alfa

INTERVENTIONS:
Drug: Recombinant human erythropoietin — Dose, route and schedule was kept same as previous erythropoietin dose at randomization; adjusted as necessary (+/- 25% of the starting dose) to maintain Hb within 11 - 12 g/dL.
  Arms: Erythropoietin
Drug: Darbepoetin Alfa — Dose conversion (100U erythropoietin = 0.42 mcg darbeopoetin). DA dose was kept once weekly (QW) if previously receiving rHuEpo ≥2 times a week, or Q2W if previously receiving rHuEpo <2 times a week. Dose was adjusted as necessary (+/- 25% of the starting dose) to maintain Hb within 11 - 12 g/dL.
  Arms: Darbepoetin alfa

SUMMARY:
The present study was designed to determine whether or not darbepoetin alfa is non-inferior to recombinant human erythropoietin in the treatment of anemia in children with chronic kidney disease stage 3-5 (on or not on dialysis).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To demonstrate that Darbepoetin alpha is non-inferior to erythropoietin for the treatment of anemia in subjects with chronic kidney disease (CKD) stage 3-5 (on or not on dialysis).

SECONDARY OBJECTIVE:

To determine the safety and tolerability of Darbepoetin alpha in the treatment of anemia in the pediatric population with CKD stage 3-5.

STUDY DESIGN:

An open-label, randomized, non-inferiority study of darbepoetin alpha (DA) and recombinant human erythropoietin(rHuEpo) for the treatment of anemia in children with chronic kidney disease stages 3 to 5 (on or not on dialysis)

DURATION OF STUDY:

The study was conducted over a period of 1 year (from 1st February 2018 to 31st January 2019).

STUDY SETTING:

This study was conducted in the Division of Pediatric Nephrology, Department of Paediatrics, Institute of Child Health, Sir Ganga Ram Hospital, New Delhi, India.

CONSENT:

A prior written informed consent was obtained from parents/ legal guardians of eligible children for participation in the study.

SAMPLE SIZE CALCULATION:

The primary objective of the study is to assess the non-inferiority of darbepoetin alfa compared with rHuEpo. Using a previous study with similar protocol [1], considering darbepoetin alfa and rHuEpo as equipotent, we accepted a type I error of 0.05 and a type II error of 0.80 for detecting a true difference. A 1.0 or greater difference in mean change in Hb variable between two groups was considered clinically significant. An estimate of standard deviation in dependent variables was assumed as 1.5. As a result, we have calculated that minimum of 28 patients are needed in each group (total-56) in order to obtain 5% type 1 error and a 80% power of detecting a difference of 1.0 or more. However, due to time constraints a sample of minimum 15 subjects in each group was planned.

Note: Sample size estimation was done by powerandsamplesize.com.

METHODOLOGY:

The study was conducted in the following phases:

1. Screening Phase (Visit 1, Day -14 to Day -1) The potential subjects were screened as per the inclusion and exclusion criteria only after obtaining written informed consent from the parent/subject.
2. Enrollment and Randomization Phase (Visit 2, Day 0)

   Subjects were randomized in two groups in a 1:1 ratio by computer generated mechanism (graphpad.com) as follows:
   1. Treatment arm 1: Erythropoietin
   2. Treatment arm 2: Darbepoetin alfa
3. Treatment Phase (Visit 3, Day 1 to Visit 8, Day 168) Patients received respective treatments for 24 week period and they were followed up every 4 weeks. Both rHuEpo and darbepoetin alfa were titrated over the first 23 weeks of the study to maintain the subjects' Hb levels between 11 to 12 g/dl without adjusting the dosing frequency. Route of administration was subcutaneous. Efficacy was determined between weeks 24 and 28.

ETHICS APPROVAL The study was approved by the Institutional Ethics Committee of Sir Ganga Ram Hospital, New Delhi.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1-18 years.
2. CKD patients stages 3 to 5 (on or not on dialysis).
3. Baseline hemoglobin 9 - 12 g/dL.
4. Subject should have adequate transferrin saturation (≥20%) and serum ferritin (≥100 ng/mL).
5. Stable erythropoietin therapy for 8 weeks ( defined as a ≤25% change in prescribed dose, no change in the route of administration and no more than one missed or withheld dose).

Exclusion Criteria:

1. Subject scheduled for a living-related kidney transplant.
2. Subject with uncontrolled hypertension.
3. HIV positive patient.
4. The patient with known hematologic disease or cause of anemia other than renal disease.
5. Patient with a history of seizure disorder or received antiepileptic medication for a seizure disorder within 6 months prior to enrolment.
6. Hyperparathyroidism (Intact parathyroid hormone more than 1500 pg/ml or biopsy proven marrow fibrosis).
7. Major surgery within 12 weeks.
8. Active inflammatory disease within 8 weeks of randomization requiring immunosuppressive therapy.
9. Clinical evidence of malignancy.
10. Blood transfusion within 8 weeks prior to initiation of therapy.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Mean change in hemoglobin (Hb) between baseline and the evaluation period | 24 -28 week
  Hb in mg/dL

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events in both groups during study period | 0-28 week

CONTACTS AND LOCATIONS:
Overall Officials: Rufaida Mazahir, MD, FNB, Principal Investigator — Sir Ganga Ram Hospital
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No
The IPD might be shared if requested from the sponsor-investigator.

REFERENCES:
- [Background] Warady BA, Arar MY, Lerner G, Nakanishi AM, Stehman-Breen C. Darbepoetin alfa for the treatment of anemia in pediatric patients with chronic kidney disease. Pediatr Nephrol. 2006 Aug;21(8):1144-52. doi: 10.1007/s00467-006-0071-0. Epub 2006 May 25. PMID 16724235
- [Background] Koshy SM, Geary DF. Anemia in children with chronic kidney disease. Pediatr Nephrol. 2008 Feb;23(2):209-19. doi: 10.1007/s00467-006-0381-2. Epub 2007 Jan 24. PMID 17245602
- [Background] Klang B, Bjorvell H, Clyne N. Quality of life in predialytic uremic patients. Qual Life Res. 1996 Feb;5(1):109-16. doi: 10.1007/BF00435975. PMID 8901373
- [Background] Gerson A, Hwang W, Fiorenza J, Barth K, Kaskel F, Weiss L, Zelikovsky N, Fivush B, Furth S. Anemia and health-related quality of life in adolescents with chronic kidney disease. Am J Kidney Dis. 2004 Dec;44(6):1017-23. doi: 10.1053/j.ajkd.2004.08.024. PMID 15558522
- [Background] Mitsnefes MM, Daniels SR, Schwartz SM, Meyer RA, Khoury P, Strife CF. Severe left ventricular hypertrophy in pediatric dialysis: prevalence and predictors. Pediatr Nephrol. 2000 Sep;14(10-11):898-902. doi: 10.1007/s004670000303. PMID 10975295
- [Background] Chavers BM, Herzog CA. The spectrum of cardiovascular disease in children with predialysis chronic kidney disease. Adv Chronic Kidney Dis. 2004 Jul;11(3):319-27. doi: 10.1053/j.arrt.2004.04.002. PMID 15241746
- [Background] Pickett JL, Theberge DC, Brown WS, Schweitzer SU, Nissenson AR. Normalizing hematocrit in dialysis patients improves brain function. Am J Kidney Dis. 1999 Jun;33(6):1122-30. doi: 10.1016/S0272-6386(99)70150-2. PMID 10352201
- [Background] Pattaragarn A, Warady BA, Sabath RJ. Exercise capacity in pediatric patients with end-stage renal disease. Perit Dial Int. 2004 May-Jun;24(3):274-80. PMID 15185776
- [Background] Sietsema KE, Hiatt WR, Esler A, Adler S, Amato A, Brass EP. Clinical and demographic predictors of exercise capacity in end-stage renal disease. Am J Kidney Dis. 2002 Jan;39(1):76-85. doi: 10.1053/ajkd.2002.29884. PMID 11774105
- [Background] Xia H, Ebben J, Ma JZ, Collins AJ. Hematocrit levels and hospitalization risks in hemodialysis patients. J Am Soc Nephrol. 1999 Jun;10(6):1309-16. doi: 10.1681/ASN.V1061309. PMID 10361870
- [Background] Ma JZ, Ebben J, Xia H, Collins AJ. Hematocrit level and associated mortality in hemodialysis patients. J Am Soc Nephrol. 1999 Mar;10(3):610-9. doi: 10.1681/ASN.V103610. PMID 10073612
- [Background] Warady BA, Ho M. Morbidity and mortality in children with anemia at initiation of dialysis. Pediatr Nephrol. 2003 Oct;18(10):1055-62. doi: 10.1007/s00467-003-1214-1. Epub 2003 Jul 23. PMID 12883982
- [Background] VanDeVoorde RG, Warady BA. Management of chronic kidney disease. In: Avner ED, Harmon WE, Niaudet P, Yoshikawa N (eds). Pediatric Nephrology, 6th edn. Springer-Verlag, Berlin, 2009; 1661-92.
- [Background] Lerner G, Kale AS, Warady BA, Jabs K, Bunchman TE, Heatherington A, Olson K, Messer-Mann L, Maroni BJ. Pharmacokinetics of darbepoetin alfa in pediatric patients with chronic kidney disease. Pediatr Nephrol. 2002 Nov;17(11):933-7. doi: 10.1007/s00467-002-0932-0. Epub 2002 Sep 14. PMID 12432437
- [Derived] Mazahir R, Anand K, Pruthi PK. Comparison of darbepoetin alpha and recombinant human erythropoietin for treatment of anemia in pediatric chronic kidney disease: a non-inferiority trial from India. Eur J Pediatr. 2023 Jan;182(1):101-109. doi: 10.1007/s00431-022-04650-1. Epub 2022 Oct 11. PMID 36220980